CLINICAL TRIAL: NCT06597019
Title: Two Part (Double-blind Inclisiran Versus Placebo [Year 1] Followed by Open-label Inclisiran [Year 2]) Randomized Multicenter Study to Evaluate Safety, Tolerability and Efficacy of Inclisiran in Children (6 to Less Than 12 Years) With Heterozygous Familial Hypercholesterolemia and Elevated LDL- Cholesterol
Brief Title: Study to Evaluate Efficacy and Safety of Inclisiran in Children With Heterozygous Familial Hypercholesterolemia
Acronym: ORION-20
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKJX839C12303; 2024-514594-21 (EudraCT Number)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Familial Hypercholesterolemia - Heterozygous
Keywords: Heterozygous familial hypercholesterolemia (HeFH),; LDL-cholesterol (LDL-C),; Children,; pediatric,; small interfering ribonucleic acid (siRNA),; inclisiran,; Familial Hypercholesterolemia,; Heterozygous FH,; Hypercholesterolemia,; Lipoprotein(a),; Hyperlipidemia,; Dyslipidemia,; Heart Failure,; Cardiovascular Diseases,; Cholesterol,; Aortic Stenosis
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypercholesterolemia; Hyperlipidemias; Dyslipidemias; Heart Failure; Cardiovascular Diseases; Aortic Valve Stenosis | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel (Year 1) to single-group (Year 2)
Who Masked: Participant, Investigator
Masking Description: Masked (Year 1) to No Masking (Year 2)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Inclisiran (Experimental): Year 1 - inclisiran sodium subcutaneous injection (given at Days 1, 90, and 270) Day 360 only - placebo subcutaneous injection Year 2 - inclisiran sodium subcutaneous injection (given at Days 450 and 630)
  Interventions: Drug: Inclisiran
- Placebo (Placebo Comparator): Year 1 - placebo subcutaneous injection (given at Days 1, 90 and 270) Year 2 - inclisiran sodium subcutaneous injection (given at Days 360, 450, and 630)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Inclisiran — Inclisiran (inclisiran sodium 300 mg subcutaneous (s.c.) for participants with body weight ≥23 kg and inclisiran sodium 180 mg s.c. for participants with body weight <23 kg. The dose level is based on the participant's body weight on Day 1 (for Part 1) and Day 360 (for Part 2), respectively.
  Other Names: KJX839
  Arms: Inclisiran
Drug: Placebo — Sterile normal saline (0.9% sodium chloride in water for subcutaneous injection)
  Other Names: saline solution
  Arms: Placebo

SUMMARY:
This is a pivotal phase III study designed to evaluate safety, tolerability, and efficacy of inclisiran in children (aged 6 to <12 years) with heterozygous familial hypercholesterolemia (HeFH) and elevated low density lipoprotein cholesterol (LDLC).

DETAILED DESCRIPTION:
This is a two-part (1 year double-blind inclisiran versus placebo / 1 year open-label inclisiran) multicenter study designed to evaluate safety, tolerability, and efficacy of inclisiran in children (aged 6 to <12 years) with heterozygous familial hypercholesterolemia (HeFH) and elevated low density lipoprotein cholesterol (LDL-C) on stable standard of care background lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, 6 to <12 years of age at screening
* HeFH diagnosed either by genetic testing or on phenotypic criteria
* Fasting LDL-C >130 mg/dL (3.4 mmol/L) at screening
* For participants 8 to <12 years, on an optimal dose of statin (investigator's discretion) unless statin intolerant, with or without other lipid-lowering therapy (e.g. ezetimibe). For participants <8 years, the use of background lipid-lowering treatment is based on investigator's discretion.
* Participants on lipid-lowering therapies (such as statin and/or e.g. ezetimibe) must be on a stable dose for ≥30 days before screening with no planned medication or dose changes during study participation.

Exclusion Criteria:

* Previous treatment (within 90 days of screening) with monoclonal antibodies directed towards PCSK9
* Secondary hypercholesterolemia, e.g. hypothyroidism or nephrotic syndrome
* Homozygous familial hypercholesterolemia (HoFH)
* Body weight <16 kg at the screening and/or randomization (Day 1) visit
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained alanine aminotransferase (ALT), aspartate aminotransferase (AST) elevation >3x ULN, or total bilirubin elevation >2x ULN (except patients with Gilbert's syndrome)
* Pregnant or nursing females
* Recent and/or planned use of other investigational medicinal products or devices

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2028-03-21 (Estimated); Study Completion 2029-04-15 (Estimated)

PRIMARY OUTCOMES:
Percentage change in LDL-C from baseline to Day 330 (Year 1) | Baseline and Day 330
  Demonstrate superiority of inclisiran compared to placebo in reducing LDL-C [percent change] at Day 330

SECONDARY OUTCOMES:
Time-adjusted percent change in LDL-C from baseline after Day 90 and up to Day 330 (Year 1) | Baseline, after Day 90 up to Day 330
  Demonstrate superiority of inclisiran compared to placebo in reducing LDL-C [time-adjusted percent change] over Year 1
Absolute change in LDL-C from baseline to Day 330 (Year 1) | Baseline and Day 330
  Demonstrate superiority of inclisiran compared to placebo in reducing LDL-C [absolute change] at Day 330 (Year 1)
Percent change in PCSK9 from baseline to Day 330 (Year 1) | Baseline and Day 330
  Demonstrate superiority of inclisiran compared to placebo in reducing PCSK9, total cholesterol, Apo B, and non-HDL-C [percent change] at Day 330 (Year 1)
Percent change in total cholesterol, non-HDL-C from baseline to Day 330 (Year 1) | Baseline and Day 330
  Demonstrate superiority of inclisiran compared to placebo in reducing PCSK9, total cholesterol, Apo B, and non-HDL-C [percent change] at Day 330 (Year 1)
Percent change in Apo B from baseline to Day 330 (Year 1) | Baseline and Day 330
  Demonstrate superiority of inclisiran compared to placebo in reducing PCSK9, total cholesterol, Apo B, and non-HDL-C [percent change] at Day 330 (Year 1)
Percent change in LDLC, total cholesterol, non-HDLC, triglycerides, HDL-C, VLDL-C from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Percent change in PCSK9 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Percent change in Apo B, Apo A1 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in LDLC, total cholesterol, non-HDLC, triglycerides, HDL-C, VLDL-C from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in PCSK9 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in Apo B, Apo A1 from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Percent change in Lp(a) from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time
Absolute change in Lp(a) from baseline to each assessment time up to Day 720 (Year 2) | Baseline, up to Day 720
  Evaluate the effect of inclisiran, compared to placebo (for Year 1) and long-term (up to Day 720), on lowering LDL-C, other lipoprotein and lipid parameters, and PCSK9 over time

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (60):
- United States (8):
  - UC San Francisco Medical Center, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Childrens National Hospital, Washington D.C., District of Columbia
  - Excel Medical Clinical Trials LLC, Boca Raton, Florida
  - Icahn School of Med at Mt Sinai, New York, New York
  - Primary Childrens Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - West Virginia Childrens Hospital, Morgantown, West Virginia
- Argentina (2):
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, CABA
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
- Brazil (4):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- China (2):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Shanghai
- Novartis Investigative Site, Prague, Czechia
- France (3):
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Hanover
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Ioannina
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Budapest, Hungary
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (4):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
- Novartis Investigative Site, Kuala Lumpur, Kuala Lumpur, Malaysia
- Novartis Investigative Site, Amsterdam, North Holland, Netherlands
- Poland (3):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz, Łódź Voivodeship
- Portugal (3):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Bloemfontein, Free State, South Africa
- Spain (8):
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Cadiz, Andalusia
  - Novartis Investigative Site, Esplugues, Barcelona
  - Novartis Investigative Site, Badalona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Seville
- Novartis Investigative Site, Taipei, Taiwan
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana, Saricam
  - Novartis Investigative Site, Ankara, Yenimahalle
  - Novartis Investigative Site, Izmir
- United Kingdom (2):
  - Novartis Investigative Site, West Midlands, Birmingham
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.